CLINICAL TRIAL: NCT00121615
Title: An Open-Label, Long-Term Extension Study to Assess the Safety and Efficacy of Etanercept in the Treatment of Psoriasis in Adult Subjects
Brief Title: Study of Etanercept in the Treatment of Psoriasis in Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040216
Record Dates: First submitted 2005-06-30; First posted 2005-07-21 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Inflammation; Psoriasis
Keywords: Clinical Trials
MeSH Terms: conditions — Inflammation; Psoriasis | interventions — Etanercept

INTERVENTIONS:
Drug: etanercept

SUMMARY:
The objective of the study is to describe the safety, tolerability, and efficacy of the long-term administration of etanercept in adults with psoriasis who have completed etanercept psoriasis study 20030115 or 20030117, in Canada, and are continuing in a long-term extension. Subjects from the 20030115 study will be followed for 24 months which began in Oct. 2004. Subjects in the 20030117 study will be followed for 12 months which began in mid 2005.

ELIGIBILITY:
Inclusion Criteria: - Subjects who completed study 20030115 or 20030117 qualify to enroll into this study (provided that they meet all inclusion/exclusion criteria). - Heterosexually active men and women of child-bearing potential must agree to use a medically acceptable form of contraception throughout the study. - Subject or designee must have the ability to self-inject investigational product. - Subject must be capable of understanding and giving written voluntary informed consent. - Negative serum pregnancy test less than or equal to 14 days prior to the first dose of investigational product in all female subjects (except those surgically sterile or at least 5 years postmenopausal) Exclusion Criteria: - Active guttate, erythrodermic, or pustular psoriasis at the time of the baseline visit - Any adverse event or infection at the time of the baseline visit or at any time during the previous etanercept psoriasis study which, in the opinion of Amgen or the Investigator, would preclude participation in the study - Presence of a serious infection less than or equal to 30 days prior to the baseline visit - Evidence of skin conditions at the baseline visit (e.g., eczema) that would interfere with evaluations of the effect of investigational product on psoriasis - Previous receipt of anti-TNF agent(s) other than etanercept - Receipt of any investigational product(s), other than etanercept, less than or equal to 30 days prior to first dose of investigational product in this study - Receipt of anti-CD4 or diphtheria IL-2 fusion protein less than or equal to 24 weeks prior to first dose of investigational product in this study - Psoralen and ultraviolet A (PUVA) light therapy less than or equal to 14 days prior to first dose of investigational product in this study - Ultraviolet A (UVA) light therapy less than or equal to 14 days prior to first dose of investigational product in this study - Ultraviolet B (UVB) light therapy less than or equal to 14 days prior to first dose of investigational product in this study - Receipt of any other systemic psoriasis therapy or oral or parenteral corticosteroids less than or equal to 14 days prior to first dose of investigational product in this study - Pregnant or breast-feeding females - Significant concurrent medical conditions prior to enrollment, including: uncontrolled hypertension (defined as systolic blood pressure measurement of greater than 180 mm Hg or an untreated diastolic blood pressure of greater than 110 mm Hg); myocardial infarction less than or equal to 52 weeks prior to baseline visit; unstable angina pectoris; uncompensated congestive heart failure; severe pulmonary disease requiring hospitalization or supplemental oxygen therapy; diagnosis of multiple sclerosis or any other demyelinating disease; insulin-dependent diabetes mellitus; history of cancer (other than in-situ cervical cancer or resected cutaneous basal cell or squamous cell carcinoma) less than or equal to 5 years prior to administration of first dose of investigational product; open cutaneous ulcers; known human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg) or hepatitis C virus (HCV) positive; any condition that might cause this study to be detrimental to the subject, in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391
Dates: Start 2004-10

PRIMARY OUTCOMES:
Subject incidence of serious adverse events, including serious infections, non-melanoma skin cancer, and all malignancies, and all adverse events.

SECONDARY OUTCOMES:
Longitudinal changes from baseline for the Physician and Patient Global Assessments and DLQI

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Papp KA, Poulin Y, Bissonnette R, Bourcier M, Toth D, Rosoph L, Poulin-Costello M, Setterfield M, Syrotuik J. Assessment of the long-term safety and effectiveness of etanercept for the treatment of psoriasis in an adult population. J Am Acad Dermatol. 2012 Feb;66(2):e33-45. doi: 10.1016/j.jaad.2010.07.026. Epub 2010 Sep 17. PMID 20850895
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20040216.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/